CLINICAL TRIAL: NCT07022704
Title: The Influence of Doxapram Administration on Diaphragmatic Excursion in Mechanically Ventilated Patients With Chronic Obstructive Pulmonary Disease Undergoing Spontaneous Breathing Trial: a Prospective Observational Study
Brief Title: Doxapram Administration on Diaphragmatic Excursion in Mechanically Ventilated Patients With Chronic Obstructive Pulmonary Disease Undergoing Spontaneous Breathing Trial
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Other Study IDs: Doxapram in COPD
Record Dates: First submitted 2025-06-07; First posted 2025-06-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: COPD; Mechanical Ventilation; Weaning From Mechanical Ventilation
Keywords: COPD; Doxapram; Diaphragmatic excursion
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Doxapram

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Doxapram: All patients will receive doxapram during spontaneous breathing trial
  Interventions: Drug: Doxapram

INTERVENTIONS:
Drug: Doxapram — Doxapram will be given as 1.5 mg/kg will be given 10 minutes after the initiation of SBT

SUMMARY:
Researchers aim to evaluate the impact of doxapram administration on diaphragmatic excursion in chronic obstructive pulmonary disease (COPD) patients undergoing spontaneous breathing trial

DETAILED DESCRIPTION:
doxapram will be administered intravenously (IV) during spontaneous breathing trial. diaphragmatic excursion will be evaluated by an expert in respiratory muscle ultrasound

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe chronic obstructive pulmonary disease undergoing spontaneous breathing trial

Exclusion Criteria:

* Refusal Allergy to doxapram neuromuscular disorders inability to evaluate the diaphragm

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary diseases undergoing breathing trial
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-06-22 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
• Diaphragmatic excursion in mm | before and 10 minutes after doxappram

SECONDARY OUTCOMES:
Arterial blood gases | before and 10 minutes after doxapram
Respiratory rate | before and 10 minutes after doxapram

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data regarding this research will be available from the corresponding author upon reasonable request

REFERENCES:
- [Background] Helmy MA, Magdy Milad L, Osman SH, Ali MA, Hasanin A. Diaphragmatic excursion: A possible key player for predicting successful weaning in patients with severe COVID-19. Anaesth Crit Care Pain Med. 2021 Jun;40(3):100875. doi: 10.1016/j.accpm.2021.100875. Epub 2021 Apr 30. No abstract available. PMID 33940248
- [Background] Pourriat JL, Baud M, Lamberto C, Fosse JP, Cupa M. Effects of doxapram on hypercapnic response during weaning from mechanical ventilation in COPD patients. Chest. 1992 Jun;101(6):1639-43. doi: 10.1378/chest.101.6.1639. PMID 1600786
- [Background] Oikawa S, Nomura H, Nishio M, Nagata R, Hata T. Doxapram hydrochloride aggravates adrenaline-induced arrhythmias accompanied by bidirectional ventricular tachycardia. ISRN Cardiol. 2014 Jan 9;2014:212045. doi: 10.1155/2014/212045. eCollection 2014. PMID 24527224
- [Background] Rutka M, Palac M, Linek P. Diaphragmatic Mobility Loss in Subjects With Moderate to Very Severe COPD May Improve After In-Patient Pulmonary Rehabilitation. Respir Care. 2021 Feb;66(2):354. doi: 10.4187/respcare.08687. No abstract available. PMID 33514664
- [Background] Scheibe N, Sosnowski N, Pinkhasik A, Vonderbank S, Bastian A. Sonographic evaluation of diaphragmatic dysfunction in COPD patients. Int J Chron Obstruct Pulmon Dis. 2015 Sep 11;10:1925-30. doi: 10.2147/COPD.S85659. eCollection 2015. PMID 26392767